CLINICAL TRIAL: NCT00136266
Title: Adherence With Iron Sprinkles Among High-Risk Infants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CDC-NCCDPHP-MM-0835-O5/05; CDC-MM-0835-O5/05
Record Dates: First submitted 2005-08-25; First posted 2005-08-29 (Estimated); Last update posted 2016-02-03 (Estimated); Status verified 2007-09

CONDITIONS: Anemia; Iron Deficiency
Keywords: Adherence; Supplements; Iron; Iron deficiency; Anemia; Vitamins; Minerals
MeSH Terms: conditions — Anemia; Iron Deficiencies | interventions — Fumigant 93; Vitamins; Minerals

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Ferrous sulphate drops with vitamins A, D, and C
Drug: Ferrous fumarate sprinkles with vitamins and minerals

SUMMARY:
Compared with iron drops, iron sprinkles supplied for 3 months to high-risk children beginning at age 5-7 months will increase adherence and reduce the rates of anemia and iron deficiency.

DETAILED DESCRIPTION:
Iron deficiency is the most common known nutrient deficiency and cause of anemia in childhood. It is associated with numerous adverse health effects, particularly delayed mental and motor development, that may be irreversible. Despite advances of iron nutrition, the prevalence of iron deficiency remains high among low-income infants and toddlers. Previous studies suggest adherence with iron containing drops is low. Adherence to iron sprinkles among children as tested in studies in less developed countries appears high.

Comparison: Children randomized to ferrous sulfate drops will be compared with children randomized to ferrous fumarate sprinkles.

ELIGIBILITY:
Inclusion Criteria:

* Healthy infants
* Age 5-7 months
* Presenting for 6 months well-child care
* Caregiver speaks English or Spanish

Exclusion Criteria:

* Pre-existing medical conditions with potential relation to iron deficiency or anemia (e.g., hemoglobinopathies, gastrointestinal disorders resulting in malabsorption, chronic renal disease, gestational age at birth of less than 36 weeks, and HIV infection)
* Inability to speak English or Spanish
* Use of vitamin or iron supplements in the previous three months

Ages: 5 Months to 7 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 128 (Actual)
Dates: Start 2005-03; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
full adherence, use of iron supplements 6-7 days/week for 3 months

SECONDARY OUTCOMES:
iron deficiency at 9 months of age
anemia at 9 months of age

CONTACTS AND LOCATIONS:
Overall Officials: Paul L. Geltman, MD, MPH, Principal Investigator — Boston University
Locations (2):
- United States (2):
  - Whittier Street Health Center, Boston, Massachusetts
  - Boston Medical Center Pediatric Primary Care Clinic, Boston, Massachusetts

REFERENCES:
- [Result] Geltman PL, Hironaka LK, Mehta SD, Padilla P, Rodrigues P, Meyers AF, Bauchner H. Iron supplementation of low-income infants: a randomized clinical trial of adherence with ferrous fumarate sprinkles versus ferrous sulfate drops. J Pediatr. 2009 May;154(5):738-43. doi: 10.1016/j.jpeds.2008.11.003. Epub 2008 Dec 25. PMID 19111318